CLINICAL TRIAL: NCT06866483
Title: Validation and Scaling of Screening Program for Undiagnosed Myasthenia Gravis-Social Media Campaign Paired With a Self-moderated Assessment
Status: Recruiting | Type: Observational
Sponsor: ZS Associates (Industry)
Collaborators: UCB Pharma (Industry); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Ananda Vishnu Pandurangadu, MD, Senior Consultant, ZS Associates
Other Study IDs: MG-002
Record Dates: First submitted 2025-03-04; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Myasthenia Gravis; Neuromuscular Disease; Neuromuscular Manifestations
Keywords: social media; myasthenia gravis
MeSH Terms: conditions — Myasthenia Gravis; Neuromuscular Diseases; Neuromuscular Manifestations | interventions — Diagnostic Self Evaluation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with undiagnosed neuromuscular symptoms
  Interventions: Behavioral: Social media recruitment; Behavioral: Self-Assessment; Behavioral: Follow-up

INTERVENTIONS:
Behavioral: Social media recruitment — Social media users exposed to a variety of paid social media advertisements as a recruitment tool for study enrollment
Behavioral: Self-Assessment — Eligible participants are asked to complete self-administered physical tests to assess inducible fatigue of specific muscle groups
Behavioral: Follow-up — Patients triaged based on their assessed risk of MG are asked to complete recommended follow-up with a clinician to determine presence of myasthenia gravis

SUMMARY:
This study expands and validates the pilot study NCT06381284. It is a fully remote, site-less, prospective, observational study enrolling adults in the United States (excluding U.S. territories) with undiagnosed neuromuscular symptoms. The primary objective is to determine the validity of a self-assessment tool in encouraging undiagnosed participants, recruited through a social media campaign, to seek medical evaluation for suspected myasthenia gravis (MG).

DETAILED DESCRIPTION:
The pilot study (NCT06381284) demonstrated the feasibility of using social media to recruit participants with undiagnosed MG-like neuromuscular symptoms. It also successfully led to the diagnosis of myasthenia gravis (MG) in previously undiagnosed individuals. In the pilot, two assessment tools were developed by the study team: the Impact of Daily Living (IDL) Survey and the MG Physical Tests. Both tools were designed using supporting literature, accepted guidelines, and a rigorous review via a panel of practicing neurologist key opinion leaders experienced in treating patients with MG.

The pilot enrolled a small cohort of participants. This current study is expanding the targeted sample size and enrollment period with the goal of validating the self-assessment tool.

Participants with undiagnosed neuromuscular symptoms, recruited through targeted social media advertisements, will complete enrollment on our study webpage.(www.unearthrootcause.com). Consented adults without specific diagnosed neurological conditions will first be screened using the IDL survey, which assesses the presence/absence of characteristic MG symptoms and habits. Qualified participants will then complete the MG Physical Tests, following video-guided instructions to perform 10 physical tests evaluating inducible muscle fatigue. A neurologist will asynchronously review the assessment results to determine whether an in-person neurology evaluation for MG is warranted. Each participant will receive a report of the neurologist's evaluation and study results to present to their doctor. Participants will be followed for up to six months with monthly survey check-ins to track whether they sought clinical evaluation and received a confirmed MG diagnosis. During follow-up participants who self-report as MG positive (newly diagnosed MG) or MG negative (MG was ruled out by physician or through testing) will be asked to upload confirmatory medical records or undergo an interview with a study navigator.

ELIGIBILITY:
Inclusion Criteria:

* Reside within the 50 states of the United States at the time of enrollment
* Age 19 or older if reside in Nebraska or Alabama, Age 21 or older if reside in Mississippi, Age 18 years or older if reside in any other state
* Active email account
* Fluency in English (spoken / written), as demonstrated by the ability to read and sign the Informed Consent Form

Exclusion Criteria:

* Live in an overseas territory of the United States
* Inability or unwillingness to provide written informed consent
* Diagnosed myasthenia gravis, including sero-negative MG*
* Diagnosed multiple sclerosis
* Have speech impairment, eye/arm/leg weakness due to diagnosed brain cancer, or stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult participants who have undiagnosed neuromuscular symptoms
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-Assessment tool validity | 6 months from time of enrollment
  Measure the specificity and sensitivity of the Self-Assessment tool

SECONDARY OUTCOMES:
Social media engagement | Enrollment period (~4-5 months)
  Measure the engagement and cost metrics of the social media ad campaign

OTHER OUTCOMES:
Time to diagnosis | 6 months from time of enrollment
  Evaluate the time to diagnosis for any participant who has a new diagnosis of MG after completing the study

CONTACTS AND LOCATIONS:
Locations (1):
- ZS Associates, Evanston, Illinois, United States

REFERENCES:
- See also: Study enrollment webpage — https://unearthrootcause.com/